CLINICAL TRIAL: NCT06875843
Title: Project VOICES: Vocal Optimization in Children Elevating the Spectrum
Acronym: Project VOICES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jena McDaniel, Assistant professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250043
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Autism
Keywords: Autism; Language; Vocalizations; Children
MeSH Terms: conditions — Autistic Disorder; Language; Vocalization, Animal

STUDY DESIGN:
Intervention Model Description: Study Design: Single case alternating treatments design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contingent responses (Experimental): Participants engage in three conditions: (a) contingent responses, (b) contingent responses with vocal elicitation strategies, (c) non-contingent control
  Interventions: Behavioral: Contingent responses; Behavioral: Contingent responses plus vocal elicitation strategies; Behavioral: Non-contingent control

INTERVENTIONS:
Behavioral: Contingent responses — The adult systematically responds to more complex child vocalizations with more complex responses. When the child first vocalizes, the adult imitates that vocalization. The child's response determines the next adult response. If the child produces a vocalization within 3 seconds, the adult imitates the child, provides a linguistic map (i.e., puts the apparent meaning into words), and complies nonverbally with the child's apparent intent (e.g., giving item or action). If the child does not produce another vocalization within 3 seconds, the adult remains quiet until the child vocalizes again.
Behavioral: Contingent responses plus vocal elicitation strategies — The adult follows the contingent responses condition protocol with the addition of using vocal toys (e.g., echo tubes, microphones that distort voices, and microphones that amplify voices) within exciting turn-taking activities/routines (e.g., blowing bubbles, balloons, and whoopee cushions). The vocal elicitation strategies emphasize the need to help children vocalize to initiate child-adult interactions. These strategies may be especially important for children who vocalize infrequently to benefit from other intervention aspects and enhance their spoken language skills. The vocal elicitation strategies are to be used when needed, rather than being obligatory for every adult-child interaction. If the child vocalizes without a vocal elicitation prompt, the adult still responds to the vocalization
Behavioral: Non-contingent control — The adult provides non-contingent vocal responses based on audio recordings from prior contingent responses condition sessions transmitted via a wireless earpiece. Recordings from these yoked sessions control for number and type of adult vocalizations and minimize the degree of contingency between adult and child vocalizations in this condition.

SUMMARY:
Thirty percent of children with autism barely talk or do not talk at all despite years of intervention. This study aims to address this important and long-standing challenge by developing a novel intervention to increase the quantity and quality of vocalizations (i.e., sounds children make before words) and expressive language in young children with autism (aged 2 to 5 years) with minimal verbal skills. The intervention includes contingent responses to the child's vocalizations and vocal elicitation strategies. We also collect social validity information from parents about how they perceive the novel intervention.

ELIGIBILITY:
Child participants

* Inclusion criteria

  * Diagnosed with autism spectrum disorder
  * Aged 2 to 5 years old
  * Use no more than 20 words (spoken, signed, or via augmentative and alternative communication) per parent report
  * Use of < 5 different words during a 15-min communication sample
  * Use of at least one consonant (observed or reported)
  * Primary language of English
* Exclusion criteria

  * Uncorrected visual or hearing impairment
  * Evidence of severe motor impairment

Caregiver participants

• Inclusion criteria

* Have a child enrolled in the study (One caregiver per child participant is enrolled.)
* Sufficient English skills to complete surveys

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of children for whom the contingent responses with vocal elicitation strategies condition is successful for increasing quantity of vocalizations | Baseline to up to 8 weeks
  The investigators will calculate the proportion of children for whom the contingent responses with vocal elicitation strategies condition is successful based on the child producing more non-vegetative vocalizations in the contingent responses with vocal elicitation strategies condition than the non-contingent control condition.
Proportion of children for whom the contingent responses condition is successful for increasing quantity of vocalizations | Baseline to up to 8 weeks
  The investigators will calculate the proportion of children for whom the contingent responses is successful based on the child producing more non-vegetative vocalizations in the contingent responses condition than the non-contingent control condition.
Proportion of children for whom the contingent responses with vocal elicitation strategies condition provides added value for increasing quantity of vocalizations | Baseline to up to 8 weeks
  The investigators will calculate the proportion of children for whom the contingent responses is successful based on the child producing more non-vegetative vocalizations in the contingent responses with vocal elicitation strategies condition than the contingent responses condition.

SECONDARY OUTCOMES:
Proportion of children for whom the contingent responses with vocal elicitation strategies condition is successful for increasing quality of vocalizations | Baseline to up to 8 weeks
  Description: The investigators will calculate the proportion of children for whom the contingent responses with vocal elicitation strategies is successful based on the child producing more vocalizations with canonical syllables, more communicative vocalizations, or a higher diversity of key consonants used in communication acts in the contingent responses with vocal elicitation strategies condition than the non-contingent control condition.
Proportion of children for whom the contingent responses condition is successful for increasing quality of vocalizations | Baseline to up to 8 weeks
  Description: The investigators will calculate the proportion of children for whom the contingent responses is successful based on the child producing more vocalizations with canonical syllables, more communicative vocalizations, or a higher diversity of key consonants used in communication acts in the contingent responses condition than the non-contingent control condition.
Proportion of children for whom the contingent responses with vocal elicitation strategies condition provides added value for increasing quality of vocalizations | Baseline to up to 8 weeks
  Description: The investigators will calculate the proportion of children for whom the contingent responses with vocal elicitation strategies condition is successful based on the child producing more vocalizations with canonical syllables, more communicative vocalizations, or a higher diversity of key consonants used in communication acts in the contingent responses with vocal elicitation strategies condition than the contingent responses condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States